CLINICAL TRIAL: NCT02045511
Title: The Baltimore HEARS Pilot Study: Hearing Health Care Equality Through Accessible Research & Solutions
Brief Title: The Baltimore HEARS Pilot Study
Acronym: HEARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NA_00088278
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Age-related Hearing Impairment 1; Personal Communication
MeSH Terms: conditions — Age-Related Hearing Impairment 1; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Treatment Group (Experimental): Immediate treatment with Baltimore HEARS intervention
  Interventions: Behavioral: Baltimore HEARS; Device: Baltimore HEARS
- Delayed Treatment Group (Placebo Comparator): 3-month delayed treatment with Baltimore HEARS intervention
  Interventions: Behavioral: Baltimore HEARS; Device: Baltimore HEARS

INTERVENTIONS:
Behavioral: Baltimore HEARS — Tailored aural rehabilitation for participant and communication partner
Device: Baltimore HEARS — Tailored fitting and programming of a personal sound amplifier. This will be accompanied by a component of aural rehabilitation.

SUMMARY:
The primary purpose of the study is to develop and test the preliminary efficacy of a first-in-kind community-based intervention to provide affordable, accessible and effective hearing health care to low-income, minority older adults.

DETAILED DESCRIPTION:
Age-related hearing impairment is strongly associated with poorer communicative functioning and social isolation, but hearing impairment often goes undiagnosed and untreated, particularly among minority and low-income older adults. Novel interventions that translate research on social engagement, minority health, and hearing technology are needed to expand delivery of hearing health care to underserved older adults. The Baltimore Hearing Equality through Accessible Research and Solutions (HEARS) project will develop and pilot a first-in-kind community-based intervention to provide affordable, accessible, and effective hearing health care to minority and low-income older adults and their communication partners. The study will follow a mixed-methods approach that will incorporate quantitative and qualitative components throughout the formative and evaluative processes. Participants and their communication partners will be randomized to an immediate treatment group or a 3-month delayed treatment group. The investigators hypothesize that the intervention is associated with increased social engagement and communication, improved quality of life, and decreased loneliness and third-party disability in the immediate treatment compared to the delayed treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* English-speaking
* Aural-oral verbal communication as primary communication modality
* Post-lingual hearing loss
* Does not currently use a hearing amplification device or hearing aid
* Signed informed consent to participate in baseline, 1 month, and 3 month assessments
* Have a communication partner able to accompany them to all study-related appointments

Exclusion Criteria:

* Individuals who do not fulfill inclusion criteria
* Score ≤ 25 on the Montreal Cognitive Assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lin, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Weinberg Senior Living Communities, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventry IM, Weinstein BE. Identification of elderly people with hearing problems. ASHA. 1983 Jul;25(7):37-42. No abstract available. PMID 6626295
- [Background] Weinstein BE. Validity of a screening protocol for identifying elderly people with hearing problems. ASHA. 1986 May;28(5):41-5. No abstract available. PMID 3718608
- [Background] Tuley MR, Mulrow CD, Aguilar C, Velez R. A critical reevaluation of the Quantified Denver Scale of Communication Function. Ear Hear. 1990 Feb;11(1):56-61. doi: 10.1097/00003446-199002000-00011. PMID 2307305
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- See also: Description of HHIE - S measure — https://consultgeri.org/try-this/general-assessment/issue-12

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Delayed Treatment Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.9 [67.2 to 79.8] | 72.2 [69.9 to 74.2] | 70.1 [68.6 to 76.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  African American or Other | 4 | 5 | 9
Hearing screening threshold [Median (Inter-Quartile Range); unit: dB HL] | 45.8 [38.8 to 59.2] | 31.7 [30 to 43.3] | 40 [32.5 to 53.3]
HHIE-S (Hearing handicap inventory for the elderly - screening) [Median (Inter-Quartile Range); unit: units on a scale] — Measure was collected through a one-on-one interview with a trained data collector.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap
  units on a scale | 19 [14.5 to 27.5] | 20 [17 to 20] | 20 [16 to 22]
Revised Quantified Denver Scale of Communication Function (QDS) [Median (Inter-Quartile Range); unit: units on a scale] — Measure was collected through a one-on-one interview conducted by a trained data collector.
  Survey includes 5 questions, scored Strongly disagree, Slightly disagree, neither, slightly agree, or strongly agree (1, 2, 3, 4, 5)
  Scoring is from 1 (worst) to 5 (best).
  The scores from the 5 questions are summed and reported as a total score. The range for the total score is 5 (worst) to 25 (best).
  Although utilized in multiple studies, including Yueh et al., 2001, there are no numerical anchors for what would represent a clinically important difference.
  units on a scale | 16 [14 to 20.2] | 16 [12.5 to 16.5] | 16 [13.5 to 18]
Revised University of California Los Angeles (UCLA) Loneliness Scale [Median (Inter-Quartile Range); unit: units on a scale] — Measure was collected via a one-on-one interview conducted by a trained data collector.
  20-item Likert-type scale. Total score is sum of the 20 items, scores range from 20 to 80. Lower values equate to lower levels of loneliness and higher values equate to higher levels of loneliness.
  Perry et al., 1990 uses the following score ranges:
  20-34 - Low degree of loneliness 35-49 - Moderate degree of loneliness 50-64 - Moderately high degree of loneliness 65-80 - High degree of loneliness
  units on a scale | 46 [43.8 to 54] | 46 [37.5 to 55.5] | 46 [41.5 to 55.5]
Patient Health Questionnaire (PHQ) [Median (Inter-Quartile Range); unit: units on a scale] — Measure collected via one-on-one interview conducted by trained data collectors.
  Total of 9 questions, scored from 0 to 3. The score from each question are summed to a total score, which can range from 0 to 27.
  Interpretation of Total Score Total Score Depression Severity 0 No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression
  units on a scale | 9.5 [4.8 to 13.8] | 8 [3 to 8.5] | 8 [4 to 11.5]
Short Form - 36 (SF) -36 mental component (Quality of Life) [Median (Inter-Quartile Range); unit: units on a scale] — Measure collected via one-on-one interview conducted by trained data collectors.
  Standard scoring can be found at http://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html.
  Higher scores indicate better mental health functioning; U.S. population norm: M = 50.0, SD = 10.0, range = [2-74].
  units on a scale | 50.9 [38 to 57.2] | 56.6 [49.7 to 59.3] | 54.4 [41.9 to 58.6]
SF-36 physical component (Quality of Life) [Median (Inter-Quartile Range); unit: units on a scale] — Measure collected via one-on-one interview conducted by trained data collectors.
  Standard scoring can be found at http://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html.
  Higher scores indicate better physical health functioning; U.S. population norm: M = 50, SD = 9.95, range = [4-71].
  units on a scale | 41.5 [40.1 to 47] | 50.6 [47.5 to 60] | 46.3 [41.5 to 59.9]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hearing Handicap Inventory for the Elderly (HHIE)-S at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  Measure Description: Measure was collected through a one-on-one interview with a trained data collector.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | -8.5 (15.4) | 0.3 (4.5)

2. Secondary Outcome: Change From Baseline in Revised QDS at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  [1] Measure Description: Measure was collected through a one-on-one interview conducted by a trained data collector.
  Survey includes 5 questions, scored Strongly disagree, Slightly disagree, neither, slightly agree, or strongly agree (1, 2, 3, 4, 5)
  Scoring is from 1 (worst) to 5 (best). Scores were summed across each of the 5 survey questions resulting in a total range of 5 (worst) to 25 (best)
  Although utilized in multiple studies, including Yueh et al., 2001, there are no numerical anchors for what would represent a clinically important difference.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | -5.9 (6.8) | -2.1 (4.3)

3. Secondary Outcome: Change From Baseline in Revised UCLA at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  [1] Measure Description: Measure was collected via a one-on-one interview conducted by a trained data collector.
  20-item Likert-type scale. Total score is sum of the 20 items, scores range from 20 to 80. Lower values equate to lower levels of loneliness and higher values equate to higher levels of loneliness.
  Perry et al., 1990 uses the following score ranges:
  20-34 - Low degree of loneliness 35-49 - Moderate degree of loneliness 50-64 - Moderately high degree of loneliness 65-80 - High degree of loneliness
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | -2.1 (10.8) | -4 (5.2)

4. Secondary Outcome: Change From Baseline in PHQ-9 at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  [1] Measure Description: Measure collected via one-on-one interview conducted by trained data collectors.
  Total of 9 questions, scored from 0 to 3. The score from each question are summed to a total score, which can range from 0 to 27.
  Interpretation of Total Score Total Score Depression Severity 0 No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression.
  Change from baseline to 3 months was reported. An increase in the score from baseline to three months (a positive number) indicates a worsening in depression severity. A decrease in the score from baseline to three months (a negative number) indicates a reduction in depression severity.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | -4.4 (6.4) | -1 (1.7)

5. Secondary Outcome: Change From Baseline in SF-36 Mental Component at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  Data were collected via one-on-one interviews with trained data collectors.
  Standard scoring can be found at http://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html.
  Higher scores indicate better mental health functioning; U.S. population norm: M = 50.0, SD = 10.0, range = [2-74].
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | 2.1 (14.7) | 1.7 (14)

6. Secondary Outcome: Change From Baseline in SF-36 Physical Component at 3 Months
Description: Mean change, Unpooled - comparing baseline to 3 month follow-up visit
  Measure collected via one-on-one interview conducted by trained data collectors.
  Standard scoring can be found at http://www.rand.org/health/surveys_tools/mos/36-item-short-form/scoring.html.
  Higher scores indicate better physical health functioning; U.S. population norm: M = 50, SD = 9.95, range = [4-71].
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 8 | 7
units on a scale | 3.6 (5.8) | -1.3 (5.4)

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored/assessed through study completion, beginning with the study start in 2/2014 through study completion in 9/2015.
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes